CLINICAL TRIAL: NCT02614352
Title: Investigate a Pharmacokinetic Characteristics and the Safety of AG1502 in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AGCA_BE_1501
Record Dates: First submitted 2015-11-24; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — Atorvastatin; candesartan

ARMS (2):
- AG1502 (Experimental)
  Interventions: Drug: Atorvastatin + Candesartan; Drug: AG1502
- Candesartan + Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin + Candesartan; Drug: AG1502

INTERVENTIONS:
Drug: Atorvastatin + Candesartan
Drug: AG1502

SUMMARY:
Primary object : Evaluate pharmacokinetic property AG1502 and Candesartan 32mg and Atorvastatin 40mg in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy males 19 to 45 years at screening.
* BMI 18-29 kg/m2

Exclusion Criteria:

* History of cardiovascular, respiratory, hepatic, renal, neuropsychiatric, endocrine, hematologic disease
* Hypersensitivity reactions to drugs or significant hypersensitivity reactions in the history of Candesartan and Atorvastatin
* Hypotension (DBP ≤ 100 mmHg or SBP ≤ 95mmHg) and hypertension (SBP ≥ 150 mmHg or DBP ≥ 95 mmHg)
* Gastrointestinal disease affected the absorption of medications
* Genetic disease of Galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
* AST or ALT > 2 x normal range
* Total bilirubin > 2.0 mg/dl
* CK > 2 x normal range
* eGFR < 60 mL/min/1.73m2
* Subject who have drunken habitually (alcohol more than 21 units/week, 1 unit = 10 g = 12.5 mL of pure alcohol) or who are unable to quit drinking during this study
* Subject who have smoke habitually more than 10 cigarettes/day or who are unable to quit smoking during this study
* Subject who treated with any investigational drugs within 90 days before the administration of investigational drug
* Previously donate whole blood within 60 days or component blood within 30 days or transfusion within 30 days
* Subject who treated with any drug within 30 days can affect absorption, distribution, metabolism, excretion of candesartan or atorvastatin
* Subject who treated with any Rx only drug or herbal drug within 14 days and any OTC within 7 days
* History of drug abuse
* Genetic neuromuscular disorder or family history of neuromuscular disorder
* Unusual diet affected the absorption, distribution, metabolism, excretion of medications
* Subjects deemed ineligible by investigator based on other reasons

Ages: 19 Years to 45 Years | Sex: Male
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Cmax (candesartan cilexetil) | 0,0.5,1,2,3,4,5,6,8,10,12,24,48 hours
AUClast (candesartan cilexetil) | 0,0.5,1,2,3,4,5,6,8,10,12,24,48 hours
Cmax (Atorvastatin) | 0,0.25,0.5,0.75,1,1.333,1.667,2,3,4,6,8,12,24,48 hours
AUClast (Atorvastatin) | 0,0.25,0.5,0.75,1,1.333,1.667,2,3,4,6,8,12,24,48 hours